CLINICAL TRIAL: NCT01919190
Title: Assessing the Impact of EXPAREL(R) on Opioid Use and Patient Reported Outcomes When Administered by Infiltration Into the Transversus Abdominis Plane (TAP) Under Ultrasound Guidance for Prolonged Postsurgical Analgesia in Lower Abdominal Surgeries
Brief Title: EXPAREL Administered by Infiltration Into the TAP for Prolonged Postsurgical Analgesia in Lower Abdominal Surgeries
Acronym: TRANSCEND
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to reasons unrelated to safety; primary endpoint signal seen during pre-specified interim analysis.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSE402
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL (Active Comparator): EXPAREL (266mg/20 ml) with 40 mL of 0.9% normal saline for a total volume of 60 mL, 30 mL to be administered to the right TAP and 30 mL to be administered to the left TAP
  Interventions: Drug: EXPAREL
- Placebo (Sham Comparator): The placebo control will be established using a grade-2 sham, no infiltration will occur
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EXPAREL — TAP with EXPAREL
  Other Names: bupivacaine liposome injectable suspension.
  Arms: EXPAREL
Drug: Placebo — Placebo
  Other Names: Placebo using grade-2 sham, no infiltration
  Arms: Placebo

SUMMARY:
The purpose of this prospective, blinded assessor, randomized trial is to assess opioid use and patient-reported outcomes of EXPAREL as a foundation in postsurgical pain therapy in Transversus Abdominis Plane (TAP) infiltration in lower abdominal surgical procedures.

DETAILED DESCRIPTION:
The purpose of this prospective, blinded assessor, randomized trial is to assess opioid use and patient-reported outcomes of EXPAREL as a foundation in postsurgical pain therapy in Transversus Abdominis Plane (TAP) infiltration in lower abdominal surgical procedures; primary endpoint signal seen during pre-specified interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >18 years of age
* American Society of Anesthesiologists (ASA) physical status 1-3
* Undergoing either lower abdominal surgery defined as Laparoscopic Hysterectomy (female), Laparoscopic Myomectomy (female), Laparoscopic Colectomy (male/female)
* Physically and mentally able to give full informed consent to participate in this study and complete all study assessments within the timeframes required (including electronic diaries should patient be discharged prior to day 4)
* Capable of returning the diary after POD 4 by mail (preferably) or upon follow up visit.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics.
* Any patient whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful local administration of EXPAREL.
* Patients who have received any investigational drug within 30 days prior to EXPAREL administration, or planned administration of another investigational product or procedure during their participation in this study.
* Any chronic condition requiring use of opioids for treatment of a medical condition for 2 weeks or more prior to surgery.
* Confirmed pregnancy at time of enrollment or breast feeding (females of child-bearing potential).
* Patients that would constitute a contraindication to participation in the study, or cause inability to comply with the study requirements.
* Any patient with diagnosed or potential metastatic disease.
* Any condition that in the investigator's opinion might be harmed or be a poor candidate for participation in the study (such as patients requiring long acting opioids as part of the induction medications).
* Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®)
* History of suspected or known addiction to, or abuse of, illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Warnott, RN, Study Director — Pacira Pharmaceuticals, Inc
Locations (13):
- United States (13):
  - Florida Hospital, Winter Park, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC St. Margaret's Hospital, Pittsburgh, Pennsylvania
  - St. John Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL: EXPAREL (266 mg/20 mL) with 40 mL of 0.9% normal saline for a total volume of 60 mL, 30 mL to be administered to the right TAP and 30 mL to be administered to the left TAP.
  EXPAREL
- Placebo: The placebo control was established using a grade-2 sham; no infiltration occurred.
  Placebo
Period: Overall Study
Arm/Group | EXPAREL | Placebo
Started | 33 (Met eligibility criteria) | 34 (Met eligibility criteria)
Completed | 30 | 34
Not Completed | 3 | 0
Not completed — Intra-op findings, etc. | 3 | 0

BASELINE CHARACTERISTICS:
Population: Who met eligibility criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL | Placebo | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Customized [Number; unit: participants]
  Under 75 | 32 | 33 | 65
  Over 75 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption Post Surgery (Cumulative Total) Until Discharge Readiness or Post Surgery Day 4
Description: Total Opioid Consumption Post Surgery (cumulative total) Until Discharge Readiness or Post Surgery Day 4
Time Frame: From surgery through 4 days postsurgery
Measure: Mean (Standard Error); unit: Opioid consumption (mg)
Groups:
- EXPAREL: EXPAREL (266 mg/20 mL) with 40 mL of 0.9% normal saline for a total volume of 60 mL, 30 mL to be administered to the right TAP and 30 mL to be administered to the left TAP
  EXPAREL
Arm/Group | EXPAREL | Placebo
Number analyzed (Participants) | 33 | 34
Opioid consumption (mg) | 3.79 (NA) — All efforts have been made to obtain the raw data but it cannot be located and a Measure of Dispersion cannot be calculated. The analysis was performed years ago, all data available have been entered. | 3.72 (NA) — All efforts have been made to obtain the raw data but it cannot be located and a Measure of Dispersion cannot be calculated. The analysis was performed years ago, all data available have been entered.
Statistical Analysis 1: Comparison: EXPAREL vs Placebo; Test type: Superiority or Other; p > 0.8, ANCOVA

2. Primary Outcome: Overall Benefit of Analgesic Score (OBAS) at Day 3
Description: Severity of postsurgical pain, satisfaction with pain management, and impact of opioid-related symptom distress measured using the Overall Benefit of Analgesic Score (OBAS) - primary endpoint is mean difference in OBAS at Day 3. (0=minimal pain and 4=maximum imaginable pain)
Time Frame: Postsurgical day 1 through day 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | EXPAREL | Placebo
Number analyzed (Participants) | 33 | 34
units on a scale | 3.05 (0.56) | 4.63 (0.56)
Statistical Analysis 1: Comparison: EXPAREL vs Placebo; Test type: Superiority or Other; p = 0.0456, Mixed Models Analysis

3. Secondary Outcome: Extent and Degree of Anesthetic Blockade
Description: Extent and degree of anesthetic blockage measured using a 5-point sensation scale.
Time Frame: Prior to TAP, immediately postoperatively, and daily through discharge or Day 4
Population: The analysis was not conducted due to the early termination of this study.
Groups:
- EXPAREL: EXPAREL (266mg /20 mL) with 40 mL of 0.9% normal saline for a total volume of 60 mL, 30 mL to be administered to the right TAP and 30 mL to be administered to the left TAP
  EXPAREL
Arm/Group | EXPAREL | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Severity of Postsurgical Pain
Description: Severity of postsurgical pain measured using an 11-point numerical rating scale (NRS 0-10).
Time Frame: Immediately in PACU postsurgery and prior to pain medication until discharge (or Day 4)
Population: The analysis was not conducted due to the early termination of this study.
Arm/Group | EXPAREL | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Quality of Recovery
Description: Measured using the Quality of Recovery 15 questionnaire (QoR-15)
Time Frame: Daily through Post Op Day 4
Population: The analysis was not conducted due to the early termination of this study.
Arm/Group | EXPAREL | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Frequency of Patient Calls Post-discharge
Description: Frequency of patient calls post-discharge related to pain and unscheduled hospital/surgeon visits
Time Frame: Post-discharge through 4 days postsurgery
Population: The analysis was not conducted due to the early termination of this study.
Arm/Group | EXPAREL | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | EXPAREL | Placebo
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EXPAREL (N=33) | Placebo (N=34)
Postoperative anemia exacerbation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Subtherapeutic international normalized ration (INR) (Investigations) | 0 (0) | 1 (1)
Postoperative abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No